CLINICAL TRIAL: NCT01633502
Title: Effects of Advanced Mechanical Circulatory Support in Patients With ST Segment Elevation Myocardial Infarction Complicated by Cardiogenic Shock. The Danish Cardiogenic Shock Trial
Brief Title: Danish Cardiogenic Shock Trial
Acronym: DanShock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Hannover Medical School (Other); University Hospital, Bonn (Other); Jena University Hospital (Other); University Hospital Dresden (Other); Heinrich-Heine University, Duesseldorf (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Charite University, Berlin, Germany (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Wuerzburg University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Jacob Moller, Professor in Cardiology, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DanShock-01
Record Dates: First submitted 2012-06-28; First posted 2012-07-04 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cardiogenic Shock Acute; Acute Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional circulatory support (Placebo Comparator): Patients randomized to conventional circulatory support.
  Interventions: Device: Conventional circulatory support
- Impella (Active Comparator): Patients randomized to Impella CP
  Interventions: Device: Impella CP

INTERVENTIONS:
Device: Conventional circulatory support — Control group treated with conventional circulatory support and observed in intensive care unit for a minimum of 48 hrs.
  Other Names: Conventional circulatory support will be employed according to enrolling sites usual management.
  Arms: Conventional circulatory support
Device: Impella CP — Control group treated with Impella CP for a minimum of 48 hrs.
  Other Names: Impella CP, Abiomed
  Arms: Impella

SUMMARY:
Cardiogenic shock a serious complication of a heart attack (myocardial infarction). Despite rapid invasive treatment, circulatory support using positive inotropes and mechanical support with intra-aortic balloon counterpulsation (IABP), and evaluation of several new treatments during the last decade, the mortality in patients with cardiogenic shock still exceeds 50%. An alternative to current management is restoration of the volume of blood pumped by the heart (cardiac output) using a ventricular assist device. In the acute setting this is difficult but can be done using the Impella device which is a catheter-based, axial flow pump that pumps blood directly from the left ventricle into the circulation thereby restoring blood flow to the failing organs. In 2012 a more powerful Impella has been introduced that is able to deliver 3.5l/min (approximately 75% of a normal cardiac output). The hypothesis of the current study is to reduce mortality and morbidity of patients with cardiogenic shock using the Impella CP. The study will be carried out as a randomized multicenter study where eligible patients will be randomized to receive conventional circulatory support or support with the Impella device and inotropic support if needed. A total of 360 patients are planned to be enrolled, and the primary endpoint will be death.

ELIGIBILITY:
Inclusion Criteria:

1. ST segment elevation myocardial infarction of less than 36 hours' duration, confirmed by new onset ST-segment elevation, or emergency angiography demonstrating acute occlusion of coronary artery, and
2. Cardiogenic shock of less than 24 hours' duration, confirmed by:

   * peripheral signs of tissue hypoperfusion (arterial blood lactate ≥2.5mmol/l and/or SvO2 <55% with a normal PaO2) and
   * systolic blood pressure less than 100mmHg and/or need for vasopressor therapy (dopamine/ norepinephrine or epinephrine), and
3. Left ventricular ejection fraction of less than 45% visually estimated or by wall motion score index >1,6.

Exclusion Criteria:

1. Other causes of shock (hypovolemia, hemorrhage, sepsis, pulmonary embolism or anaphylaxis).
2. Shock due to mechanical complication to myocardial infarction (papillary muscle rupture, rupture of the ventricular septum or rupture of free wall).
3. Severe aorta valve regurgitation/stenosis.
4. Predominant right ventricular failure.
5. Out of hospital cardiac arrest with persistent Glasgow coma scale <8 after return of spontaneous circulation.
6. Shock duration>24 hours.
7. Known heparin intolerance.
8. Already established mechanical circulatory support
9. Do not resuscitate wish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2012-12; Primary Completion 2023-07 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Death | up to 6 months
  Death from all causes

SECONDARY OUTCOMES:
MACE | minimum follow-up 6 months
  Major cardiovascular events, death, cardiac transplant, escalation to permanent left ventricular assist device, re-hospitalization for heart failure.
Composite saftey | up to 6 months
  Combined safety comprising major bleeding, vascular complications, and significant hemolysis.
Days alive out of hospital | up tp 6 months
  Days alive and out of hospital; calculated by subtracting the number of days spent in hospital, from time of randomization to end of follow-up (180 days) for each patient.

OTHER OUTCOMES:
Hemodynamics | up to 7 days
  Cardiac power index
Hemodynamics | up to 7 days
  Lactate clearence
Hemodynamics | up to 7 days
  Pulmonary artery pulsatility index
Health economics | up to 6 months
  Cost of treatments
Renal function | up to 30 days
  Development of acute kidney injury and need for dialysis
Bleeding | up to 30 days
  Bleeding complications during admission
Revascularization strategy | During procedure
  Syntax score ( a grading system that evaluates the complexity and prognosis of patients undergoing percutaneous coronary intervention, higher scores denotes more complex disase and higher risk)
Revascularization strategy | up to 6 months
  Additional non culprit revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Jacob E Moller, MD, Principal Investigator — Department of Cardiology, Odense University Hospital, Odense; Anders Junker, MD, Study Chair — Department of Cardiology, Odense University Hospital; Christian Hassager, MD, Study Chair — Department of Cardiology, Copenhagen University Hospital Gentofte; Andreas Shaefer, MD, Study Chair — Hannover Medical School; Nikos Werner, MD, Study Chair — University Hospital Trier
Locations (13):
- Denmark (3):
  - Aarhus University Hospital Skejby, Aarhus
  - Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- Germany (9):
  - Charite Berlin, Berlin
  - University Hospital Bonn, Bonn
  - Dresden University Hospital, Dresden
  - Düsseldorf University Hospital, Düsseldorf
  - UKE Hamburg, Hamburg
  - Hannover Medical School, Hanover
  - Jena University Hospital, Jena
  - Brüderkrankenhaus Trier, Trier
  - University Hospital Würzburg, Würzburg
- NHs Harefield Hospital, London, United Kingdom

REFERENCES:
- [Background] Moller JE, Gerke O; DanGer Shock Investigators. Danish-German cardiogenic shock trial-DanGer shock: Trial design update. Am Heart J. 2023 Jan;255:90-93. doi: 10.1016/j.ahj.2022.10.078. Epub 2022 Oct 19. PMID 36272450
- [Background] Udesen NJ, Moller JE, Lindholm MG, Eiskjaer H, Schafer A, Werner N, Holmvang L, Terkelsen CJ, Jensen LO, Junker A, Schmidt H, Wachtell K, Thiele H, Engstrom T, Hassager C; DanGer Shock investigators. Rationale and design of DanGer shock: Danish-German cardiogenic shock trial. Am Heart J. 2019 Aug;214:60-68. doi: 10.1016/j.ahj.2019.04.019. Epub 2019 May 6. PMID 31176289
- [Result] Moller JE, Engstrom T, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Frydland M, Holmvang L, Kjaergaard J, Sorensen R, Lonborg J, Lindholm MG, Udesen NLJ, Junker A, Schmidt H, Terkelsen CJ, Christensen S, Christiansen EH, Linke A, Woitek FJ, Westenfeld R, Mobius-Winkler S, Wachtell K, Ravn HB, Lassen JF, Boesgaard S, Gerke O, Hassager C; DanGer Shock Investigators. Microaxial Flow Pump or Standard Care in Infarct-Related Cardiogenic Shock. N Engl J Med. 2024 Apr 18;390(15):1382-1393. doi: 10.1056/NEJMoa2312572. Epub 2024 Apr 7. PMID 38587239
- [Derived] Jensen LO, Beske RP, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Holmvang L, Wachtell K, Engstom T, Udesen NLJ, Schmidt H, Junker A, Terkelsen CJ, Christensen S, Linke A, Moller JE, Hassager C; DanGer Shock Investigators. Delay From First Symptoms in Patients Presenting With STEMI and Cardiogenic Shock: Insights From the DanGer Shock Trial. Circ Cardiovasc Interv. 2026 Jan 12:e015718. doi: 10.1161/CIRCINTERVENTIONS.125.015718. Online ahead of print. PMID 41521915
- [Derived] Mangner N, Beske RP, Hassager C, Jensen LO, Eiskjaer H, Linke A, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Engstrom T, Holmvang L, Lonborg JT, Udesen NLJ, Schmidt H, Junker A, Terkelsen CJ, Schrage B, Woitek FJ, Moller JE; DanGer Shock Investigators. Sex-Specific Microaxial Flow Pump Use and Outcomes in Infarct-Related Cardiogenic Shock in the DanGer Shock Trial. J Am Coll Cardiol. 2025 Oct 17:S0735-1097(25)07782-4. doi: 10.1016/j.jacc.2025.09.019. Online ahead of print. PMID 41222528
- [Derived] Mikkelsen AD, Beske RP, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze C, Skurk C, Nordbeck P, Schrage B, Panoulas V, Zimmer S, Schafer A, Engstrom T, Holmvang L, Frydland M, Junker AB, Schmidt H, Udesen NLJ, Wachtell K, Terkelsen CJ, Linke A, Kjaergaard J, Moller JE, Hassager C; DanGer Shock Investigators. Systolic Blood Pressure and Microaxial Flow Pump-Associated Survival in Infarct-Related Cardiogenic Shock: A Post Hoc Analysis of the DanGer Shock Randomized Clinical Trial. JAMA Cardiol. 2025 Nov 1;10(11):1157-1165. doi: 10.1001/jamacardio.2025.3337. PMID 40884241
- [Derived] Moller JE, Beske RP, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Schrage B, Panoulas V, Zimmer S, Schafer A, Werner N, Holmvang L, Kjaergaard J, Engstom T, Udesen NLJ, Schmidt H, Junker A, Wachtell K, Terkelsen CJ, Christensen S, Linke A, Burkhoff D, Hassager C; DanGer Shock Investigators. Effect of Microaxial Flow Pump on Hemodynamics in STEMI-Related Cardiogenic Shock. J Am Coll Cardiol. 2025 Jul 1;85(25):2456-2468. doi: 10.1016/j.jacc.2025.04.062. PMID 40562510
- [Derived] Klein A, Beske RP, Hassager C, Jensen LO, Eiskjaer H, Mangner N, Linke A, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Engstom T, Holmvang L, Junker A, Schmidt H, Terkelsen CJ, Moller JE; DanGer Shock Investigators. Treating Older Patients in Cardiogenic Shock With a Microaxial Flow Pump: Is it DANGERous? J Am Coll Cardiol. 2025 Feb 18;85(6):595-603. doi: 10.1016/j.jacc.2024.11.003. Epub 2024 Nov 15. PMID 39551167
- [Derived] Zweck E, Hassager C, Beske RP, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Kelm M, Engstrom T, Holmvang L, Junker A, Schmidt H, Terkelsen CJ, Linke A, Westenfeld R, Moller JE; DanGer Shock Investigators. Microaxial Flow Pump Use and Renal Outcomes in Infarct-Related Cardiogenic Shock: A Secondary Analysis of the DanGer Shock Trial. Circulation. 2024 Dec 17;150(25):1990-2003. doi: 10.1161/CIRCULATIONAHA.124.072370. Epub 2024 Oct 27. PMID 39462276
- [Derived] Udesen NLJ, Beske RP, Hassager C, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Frydland M, Holmvang L, Kjaergaard J, Engstom T, Schmidt H, Junker A, Terkelsen CJ, Christensen S, Linke A, Moller JE; DanGer Shock Investigators. Microaxial Flow Pump Hemodynamic and Metabolic Effects in Infarct-Related Cardiogenic Shock: A Substudy of the DanGer Shock Randomized Clinical Trial. JAMA Cardiol. 2025 Jan 1;10(1):9-16. doi: 10.1001/jamacardio.2024.4197. PMID 39462240